CLINICAL TRIAL: NCT05605054
Title: An RCT Testing a Health Literacy Intervention to Reduce Disparities in Access to Care Among Minority Justice-Involved Adults
Brief Title: UCSD RELINK: Connecting Adults To Supportive Services
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Victoria D. Ojeda (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor-Investigator, Victoria D. Ojeda, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 161903; R01MD016959 (NIH)
Record Dates: First submitted 2022-10-11; First posted 2022-11-04 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Health Care Utilization
Keywords: Justice Involved Adults; Re-entry Population; Health Coaching; Service Navigation
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coach-guided (Experimental): In person or phone call with an assigned Health Coach for about 1 hour per week for 12 weeks to complete the Health Literacy course, and with an assigned Service Navigator for 30 minutes per week for 12 weeks to address health and social service needs.
  Interventions: Behavioral: UCSD RELINK
- Self study (Active Comparator): Self-guided printed or online version of the Health Literacy course (approximately 1 hour per week for 12 weeks) and comprehensive Service Navigation report with recommended referrals to services, providers, and contact information for service providers so that the participant can access these resources independently (i.e., without Navigator assistance).
  Interventions: Behavioral: Self-study

INTERVENTIONS:
Behavioral: UCSD RELINK — UCSD RELINK coach-guided health literacy intervention and in-person service navigation assistance
  Arms: Coach-guided
Behavioral: Self-study — Self-studying of programmatic information and list of service referrals
  Arms: Self study

SUMMARY:
The goal of this randomized intervention study is to learn about effective health literacy teaching methods in Justice Involved Adults (JIA).

Researchers will compare coach-guided health literacy or self-study design to see if there is a difference in the access and use of healthcare in this population.

The main questions it aims to answer are:

* Will this improve access and use of heath services?
* Will this improve health insurance coverage and long term use of health services?

Participants will:

* Meet with a health coach and service navigator during 12 sessions or meet with service navigator and complete online training over 12 weeks.
* Complete surveys at different time (6months, 1 year)

DETAILED DESCRIPTION:
Health literacy refers to the skills needed to effectively access, understand, and use health resources. Inadequate health literacy annually costs the U.S. $100-$200 billion and is observed among justice involved adults (JIA)-a group of ~20 million U.S. persons who are disproportionately non-elderly and African American, Black, and Hispanic due to systemic racism and over-policing. JIA face numerous barriers in accessing healthcare which contributes to a high, lifelong burden of chronic and infectious disease. Healthcare access is defined as 1) having health insurance coverage, 2) having a regular source of care and 3) obtaining healthcare in a timely manner. Health literacy interventions for JIA are critically needed but are unavailable and NIH-funded research that is inclusive of JIA is sorely lacking. This timely study addresses these gaps. This study will implement a longitudinal mixed-methods randomized clinical trial (RCT) to assess the impact of the UCSD RELINK coach-guided health literacy intervention vs. a self-study control group on JIA's healthcare access. To achieve this aim, 300 JIA ages 18+ will be recruited in San Diego, CA and randomized 1:1 to the Treatment Group (i.e., coach-guided health literacy intervention) or the Control Group (i.e., self-study of the intervention). This study is timely and may inform health literacy interventions for JIA, policies to build health literacy among JIA in institutional and community settings, and the service delivery models for JIA. The proposed intervention has great potential for increasing health literacy among JIA and thus improving the well-being of this sizeable and underserved community. Findings from this study may also have relevance for interventions seeking to build the health literacy of other low-income communities.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Persons, aged 18 and over
4. Resident of San Diego County
5. Not incarcerated at time of enrollment
6. Justice involved in the past 3 years (on parole, probation, court diverted)
7. Understands English
8. Access to a cell phone

Exclusion Criteria:

1. Under the age of 18 years old
2. Not a resident of San Diego County
3. Incarcerated at enrollment
4. Not justice-involved within the last 3 years (i.e., not on probation or parole or was court-diverted in the past 3 years)
5. No access to a cell phone
6. Cannot provide informed consent
7. Does not understand English
8. Previously enrolled in the pilot UCSD RELINK program
9. Adults who have current or prior convictions related to sexual violence/abuse (Penal Code [PC] 290), lewd acts with a child (PC 288), child abduction (PC 280), or arson (PC 451)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Recent Use of Health Services | 6 months
  Any healthcare use in the past 6 months (vs. never received services or received services more than 6 months ago)

SECONDARY OUTCOMES:
Health Insurance Coverage | 6 months
  Defined as uninsured versus any insurance
Regular Source of Care | 6 months
  Presence of one (or multiple) source(s) of care identified by participants

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Ojeda, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - Center for employment opportunities, San Diego, California
  - San Diego Probation Department, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ojeda VD, Berliant E, Parker T, Lyles M, Edwards TM, Jimenez C, Linke S, Hiller-Venegas S, Lister Z. Overview of a Pilot Health-focused Reentry Program for Racial/Ethnic Minority Probationers ages 18 to 26 in Southern California. Int J Offender Ther Comp Criminol. 2022 Sep;66(12):1303-1326. doi: 10.1177/0306624X211013739. Epub 2021 May 12. PMID 33980068